CLINICAL TRIAL: NCT00994006
Title: The Absorption of Supplemental Magnesium Oxide Compared to Magnesium Citrate in Healthy Subjects With no Apparent Heart Disease
Brief Title: The Absorption of Magnesium Oxide Compared to Citrate in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Michael Shechter, MD, MA, PI, Leviev Heart Center, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-7339-09-SMC
Record Dates: First submitted 2009-10-11; First posted 2009-10-14 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Subjects; Hypomagnesemia
Keywords: Magnesium; nutrition; platelets; aggregation
MeSH Terms: interventions — Magnesium Oxide; magnesium citrate; levulinic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium oxide tables (Active Comparator): Subjects will be instructed to take Magnox 520 qd
  Interventions: Dietary Supplement: Magnesium oxide
- Magnesium citrate tablets (Active Comparator): Subjects will be instructed to take magnesium diasporal tablets t.i.d.
  Interventions: Dietary Supplement: Magnesium citrate

INTERVENTIONS:
Dietary Supplement: Magnesium oxide — 520 mg of elemental magnesium q.d.
  Other Names: Magnox 520 TM
  Arms: Magnesium oxide tables
Dietary Supplement: Magnesium citrate — Magnesium citrate , 98.6 mg of elemental magnesium t.i.d.
  Other Names: Magnesium Diasporal
  Arms: Magnesium citrate tablets

SUMMARY:
The magnesium food content in the Western world is consistently reducing. Hypomagnesemia is common in hospitalized patients, especially in the elderly with coronary artery disease (CAD) and/or those with chronic heart failure. Hypomagnesemia is associated with increased incidence of diabetes mellitus, metabolic syndrome, mortality rate from coronary artery disease (CAD) and all cause. Magnesium supplementation improves myocardial metabolism, inhibits calcium accumulation and myocardial cell death; it improves vascular tone, peripheral vascular resistance, afterload and cardiac output, reduces cardiac arrhythmias and improves lipid metabolism. Magnesium also reduces vulnerability to oxygen-derived free radicals, improves human endothelial function and inhibits platelet function, including platelet aggregation and adhesion. The data regarding the absorption difference between supplemental magnesium oxide and magnesium citrate in humans is spare.

DETAILED DESCRIPTION:
Two oral preparations of magnesium are available in Israel:

1. Magnesium Diasporal (magnesium citrate, elemental magnesium 98.6 mg), PROTINA GMBH, ISMANING, Germany
2. Magnox 520 TM (magnesium oxide, 520 mg elemental magnesium), Naveh Pharma Ltd., Israel.

The data regarding the absorption difference between the two supplemental magnesium preparations (magnesium oxide and magnesium citrate) in humans is spare.

Primary objective: To find out the absorption of magnesium citrate compared to magnesium oxide in healthy subjects with no apparent heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-70 years
2. Healthy subjects

Exclusion Criteria:

1. Chest pain
2. Diabetes mellitus
3. Documented coronary artery disease
4. Asthma or any lung disease
5. Chronic diarrhea
6. Chronic renal failure (serum creatinine> 3 mg/dL)
7. Hypo or hyperthyroidism
8. Heart failure
9. On any chronic therapy/medications
10. Malabsorption
11. AV block
12. Pacemaker
13. Any malignancy
14. Obesity > 30 kg/m2 body mass index
15. Smokers
16. Pregnancy
17. Alcohol or drug abuse
18. Any chronic inflammation
19. Refuse to sign inform consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Intracellular magnesium levels will be assessed | 30-day

SECONDARY OUTCOMES:
Platelet function tests | 30-day

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, MA, Principal Investigator — The Leviev Heart Center, Sheba Medical Center
Locations (1):
- The Leviev Heart Center, Chaim Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel

REFERENCES:
- [Background] Shechter M. Magnesium and cardiovascular system. Magnes Res. 2010 Jun;23(2):60-72. doi: 10.1684/mrh.2010.0202. Epub 2010 Mar 31. PMID 20353903
- [Derived] Shechter M, Saad T, Shechter A, Koren-Morag N, Silver BB, Matetzky S. Comparison of magnesium status using X-ray dispersion analysis following magnesium oxide and magnesium citrate treatment of healthy subjects. Magnes Res. 2012 Mar 1;25(1):28-39. doi: 10.1684/mrh.2012.0305. PMID 22433473